CLINICAL TRIAL: NCT01424371
Title: A Case-Control Study to Evaluate the Effectiveness of Adjuvanted Trivalent Inactivated Influenza Vaccine in the Elderly Aged ≥65 Years.
Brief Title: Adjuvanted Influenza Vaccine Effectiveness in the Elderly (65+Yrs)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fraser Health (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Paul VanBuynder, Chief Medical Health Officer, Fraser Health
Other Study IDs: 2011-071
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adjuvanted Vaccine Group
- Unadjuvanted Vaccine Group
- Unvaccinated Elderly

SUMMARY:
This study explores the hypothesis that the use of an adjuvanted influenza vaccine in the elderly will produce greater vaccine effectiveness in their group.

DETAILED DESCRIPTION:
To evaluate the effectiveness of adjuvanted trivalent inactivated influenza vaccine in the elderly (aged ≥ 65 years) through the reduction in relative risk of microbiologically confirmed influenza illness

ELIGIBILITY:
Inclusion Criteria:

1.Elderly tested for influenza as part of routine clinical care in the Lower Mainland and on Vancouver Island during the influenza season.

Cases: Proven influenza diagnosed on naso-pharyngeal swab via PCR Controls: Elderly with influenza-like-illness testing negative for influenza during the influenza season.

Exclusion Criteria:

1. Known immunodeficiency disorders (including HIV)
2. Current or recent (within 90 days prior to first dose of influenza vaccine) immunosuppressive treatment including chronic oral steroids (1mg/kg for > 4 weeks), cytotoxic chemotherapy, radiation therapy, other immunosuppressive drug and biologic agents Note: Use of topical or inhalant corticosteroids is acceptable.
3. Administration of immunoglobulins during the study period;

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All elderly over 65 years in the lower mainland of British Columbia presenting with an influenza-like-illness
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Vaccine effectiveness against laboratory confirmed influenza illness | Influenza season 2011/12 and 2012/13
  Evaluation of the effectiveness of an adjuvanted TIV in the elderly aged ≥65 years, through the reduction in relative risk of microbiologically confirmed influenza illness

CONTACTS AND LOCATIONS:
Overall Officials: PAUL G VAN BUYNDER, MBBS MPH, Principal Investigator — Fraser Health Authority
Locations (1):
- Fraser Health Authority, Surrey, British Columbia, Canada